CLINICAL TRIAL: NCT07262905
Title: Sedation Related Respiratory Deterioration in COPD: Risk Indicators and Predictive Performance of the Integrated Pulmonary Index
Brief Title: Risk Indicators and IPI Performance in Sedation-Related Respiratory Deterioration in COPD
Acronym: IPI-COPD
Status: Completed | Type: Observational
Sponsor: Umran Karaca (Other Government)
Responsible Party: Sponsor-Investigator, Umran Karaca, Assoc. Prof. of Anesthesiology and Reanimation, Bursa Yuksek Ihtisas Training and Research Hospital
Organization: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Other Study IDs: BursaYIERH-05; 2024-TBEK 2025/01-13 (Other: Bursa Yuksek Ihtisas Training and Research Hospital, Ethics Committee)
Record Dates: First submitted 2025-11-16; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Endoscopy, Gastrointestinal
Keywords: COPD, Integrated Pulmonary Index, capnography, sedation, endoscopy, hypoventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypoventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD Cohort: This cohort includes patients with chronic obstructive pulmonary disease (COPD) undergoing combined gastroscopy and colonoscopy under routine sedation. No study-related interventions are administered. Participants will be classified during analysis based on whether a clinical intervention becomes necessary during the procedure.
  Interventions: Other: Sedation Analgesia and Respiratory Monitoring (Integrated Pulmonary Index - IPI)

INTERVENTIONS:
Other: Sedation Analgesia and Respiratory Monitoring (Integrated Pulmonary Index - IPI) — Patients underwent routine combined gastroscopy and colonoscopy performed under standard sedation as part of usual clinical care. No study-related interventions were administered. All monitoring procedures, including the Integrated Pulmonary Index (IPI), were part of standard clinical practice.

SUMMARY:
This prospective observational clinical study investigates two key questions in COPD patients undergoing sedated endoscopic procedures. The first is whether respiratory deterioration that may occur during the procedure is associated with clinical risk indicators such as symptom burden, prior exacerbations, and previous hospitalizations. The second is to assess the effectiveness of the Integrated Pulmonary Index (IPI) in predicting this deterioration, and to compare its performance with traditional respiratory monitoring parameters including oxygen saturation (SpO₂) and capnography (EtCO₂).

The study hypothesis is that respiratory deterioration is linked to clinical risk indicators and that the IPI will demonstrate superior predictive accuracy compared with classical monitoring parameters.

All participants will belong to a single COPD cohort and will not be assigned to different intervention arms. For analysis, patients will be categorized based on whether clinical interventions-such as increased oxygen flow, repositioning, or respiratory support-become necessary during the procedure. This classification reflects routine clinical care, and no additional interventions are performed as part of the study.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a progressive disorder characterized by persistent airflow limitation, with dyspnea and productive cough being the predominant clinical features. According to the GOLD 2024 guidelines, the one-year history of exacerbations, including both the number of exacerbations and associated hospitalizations, represents the strongest predictor of future risk in COPD. The A-B-E classification system, based on symptom severity (CAT score) and exacerbation history, provides a structured framework for defining the clinical risk level of COPD patients.

Sedation in individuals with COPD can lead to rapid deterioration of respiratory function due to markedly limited ventilatory reserve. In this high-risk population, hypoventilation, apnea, desaturation, or alterations in capnographic waveforms during sedation constitute key indicators of respiratory compromise. While conventional monitoring parameters such as SpO₂, EtCO₂, respiratory rate, and pulse rate evaluate specific components of respiratory physiology individually, the Integrated Pulmonary Index (IPI) consolidates these four parameters into a single composite score reflecting both oxygenation and ventilation status. This integrated approach may facilitate earlier and more reliable detection of respiratory deterioration.

This prospective observational study focuses on two primary questions. First, it aims to investigate the relationship between respiratory deterioration occurring during sedated procedures and clinical risk indicators such as symptom severity (CAT score), the number of exacerbations in the previous year, and associated hospital admissions. Second, it seeks to evaluate the predictive performance of the IPI for identifying such respiratory deterioration and to compare its accuracy with classical respiratory monitoring parameters, namely SpO₂ and EtCO₂. This comparison will help determine whether the IPI provides an additional early-warning advantage for COPD patients undergoing sedation.

All participants will be included in a single COPD cohort, and the study involves no randomization or intervention arms. During data analysis, patients will be classified according to whether clinical interventions, such as increased oxygen supplementation, repositioning, or respiratory support, become necessary during the procedure. This classification reflects routine clinical decision-making and does not represent an intervention introduced by the study protocol.

The study hypothesizes that respiratory deterioration during sedation is associated with established clinical risk indicators and that the IPI will demonstrate higher predictive accuracy than conventional respiratory monitoring parameters.

This minimal-risk observational investigation is based solely on the assessment of standard clinical monitoring data obtained during routine sedated endoscopic procedures; no additional procedures or interventions are performed within the scope of the study.

ELIGIBILITY:
Inclusion Criteria:Age ≥ 18 years

Diagnosed with Chronic Obstructive Pulmonary Disease (COPD) according to GOLD 2024 criteria

Classified as ASA physical status I-IV

Undergoing elective gastrointestinal endoscopic procedure under sedation analgesia

Suitable for sedation outside the operating room

Provided written informed consent -

Exclusion Criteria:

Age < 18 years

Unstable cardiovascular or respiratory condition

Requirement for general anesthesia or advanced airway management

Pregnancy

Known hypersensitivity to sedative medications

Refusal or inability to provide informed consent

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with confirmed COPD undergoing elective gastrointestinal endoscopic procedures under sedation analgesia at a tertiary training and research hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Association Between Respiratory Deterioration and COPD-Specific Clinical Risk Indicators | 0, 3, 5, 10, 15, and 20 minutes during the procedure.
  Respiratory deterioration (yes/no) requiring clinical intervention during sedated combined gastroscopy-colonoscopy will be assessed for its association with baseline COPD-specific risk indicators, including the COPD Assessment Test (CAT) score, one-year exacerbation frequency, and COPD-related hospitalizations.

SECONDARY OUTCOMES:
Diagnostic Performance of the Integrated Pulmonary Index (IPI) for Predicting Respiratory Deterioration | 0, 3, 5, 10, 15, and 20 minutes during the procedure.
  The ability of the Integrated Pulmonary Index (IPI) to predict respiratory deterioration during sedated gastrointestinal endoscopy will be evaluated and compared with conventional respiratory monitoring parameters (SpO₂ and EtCO₂). Diagnostic performance will be summarized using accuracy metrics.

CONTACTS AND LOCATIONS:
Overall Officials: Füsun Gözen, MD (Anesthesiology), Principal Investigator — SBÜ Bursa Yüksek İhtisas Training and Research Hospital, University of Health Sciences (SBÜ)
Locations (1):
- Bursa Yüksek İhtisas Training and Research Hospital, Bursa, Marmara Region, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Deidentified individual participant data will not be shared due to institutional policies and lack of patient consent for data sharing.Study protocol and statistical analysis plan will be available upon reasonable request from the corresponding author.

REFERENCES:
- [Background] Karaarslan FN, Ozturk ZS, Isik GC, Cevik Y. Value of integrated pulmonary index to predict exacerbation of chronic obstructive pulmonary Disease's severity. Am J Emerg Med. 2023 Sep;71:54-58. doi: 10.1016/j.ajem.2023.05.043. Epub 2023 Jun 8. PMID 37331230